CLINICAL TRIAL: NCT03412084
Title: Translating a "Stand Up and Move More" Intervention by State Aging Units to Older Adults in Underserved Communities
Brief Title: A "Stand Up and Move More" Intervention for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-1155; R21AG054916 (NIH); A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW, Madison)
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary Lifestyle; physical function
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stand up intervention (Experimental): four week behavioral intervention based on self-regulation theory which is designed to facilitate the development of action plans to break up prolonged sitting
  Interventions: Behavioral: Stand up and move more
- Control (No Intervention): No behavioral intervention - the control group will go about their daily life, but come in for assessments at the same time points as the intervention group

INTERVENTIONS:
Behavioral: Stand up and move more — 4 week behavioral intervention involving the development and implementation of action plans
  Arms: Stand up intervention

SUMMARY:
The purpose of the expanded study is to examine the effectiveness of a "Stand Up and Move More" intervention to reduce sedentary behavior in older adults from underserved communities.

DETAILED DESCRIPTION:
Based on successful pilot research in Rock County, WI, and the receipt of funding from the National Institutes of Health, the investigators expanded research to additional counties in Wisconsin for a total of four counties (i.e., Dane, Iowa, Rock, and Vilas counties). Sample size will increase and participants will be randomly assigned to the intervention group (Stand Up and Move More group) or a wait-list control group (who receive the intervention after 12 weeks). The Stand Up and Move More intervention/workshop involves sessions once/week for four weeks with a refresher session at 8 weeks. Assessments will be conducted before the intervention/workshop begins, and then again at 4 weeks and 12 weeks. We have added several questionnaires to examine potential mediators of behavior change (e.g., self-efficacy, self-regulation, outcome expectancies).

ELIGIBILITY:
Inclusion Criteria:

* adults older than 55 yrs of age
* inactive or low active (i.e., less than 60 minutes of physical activity/week)
* residents of Dane, Iowa, Rock or Vilas counties, and
* residing in a home or an apartment.

Exclusion Criteria:

* low levels of sedentary behavior (less than or equal to 6 hours/day),
* recent hospitalization (i.e., past month),
* uncontrolled medical conditions including: uncontrolled hypertension, heart disease, actively receiving chemotherapy or palliative care for cancer, stage 4 liver disease, end-stage renal or pulmonary disease, severe arthritis or any other orthopedic condition that could be made worse by standing up and moving more;
* inability to stand up without assistance of another person, and
* inability to speak or hear spoken English.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Koltyn, PhD, Principal Investigator — UW-Madison
Locations (1):
- Kelli Koltyn, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stand up Intervention | Control
Started | 48 | 36
Completed | 44 | 35
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Participant moved | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stand up Intervention | Control | Total
Number analyzed (Participants) | 48 | 36 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9) | 73.5 (6) | 73 (8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 42 | 32 | 74
  Gender: Male | 6 | 3 | 9
  Gender: Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 23 | 60
  Unknown or Not Reported | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 31 | 25 | 56
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 48 | 36 | 84

OUTCOME MEASURES:

1. Primary Outcome: Total Sedentary Time Per Day
Description: Participants wore monitors during the day to assess total sitting time/day
Time Frame: Baseline, 4 weeks, 12 weeks
Population: The number of participants analyzed differs for each time point due to participant availability, attrition, and not all participants wore the monitors per protocol for each visit (10 hours/day for a full week each time point).
Measure: Mean (Standard Deviation); unit: minute/day
Arm/Group | Stand up Intervention | Control
Number analyzed (Participants) | 48 | 36
minute/day
  Baseline: number analyzed (Participants) | 37 | 30
  Baseline | 618 (119) | 660 (153)
  4 weeks: number analyzed (Participants) | 32 | 30
  4 weeks | 564 (119) | 650 (117)
  12 weeks: number analyzed (Participants) | 26 | 22
  12 weeks | 602 (116) | 617 (120)

2. Secondary Outcome: Short Physical Performance Battery (SPPB) Score
Description: The SPPB is an assessment of physical limitations. It combines scores from a balance test, gait speed test, and a chair stand test. The total possible range of scores is 1-12, higher scores indicate better function/less functional limitations.
Time Frame: Baseline, 4 weeks, 12 weeks
Population: The number of participants analyzed differs for each time point due to participant availability and attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stand up Intervention | Control
Number analyzed (Participants) | 48 | 36
score on a scale
  Baseline: number analyzed (Participants) | 43 | 34
  Baseline | 8.05 (2.46) | 7.65 (2.60)
  4 weeks: number analyzed (Participants) | 41 | 36
  4 weeks | 9.29 (2.65) | 7.44 (2.31)
  12 weeks: number analyzed (Participants) | 29 | 25
  12 weeks | 10.45 (2.01) | 8.00 (2.81)

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Arm/Group | Stand up Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/36
Other Adverse Events (participants affected / at risk) | 0/48 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03412084/Prot_SAP_000.pdf